CLINICAL TRIAL: NCT04675203
Title: Molecular Mechanisms of Tooth Eruption
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7946
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Tooth Eruption
MeSH Terms: conditions — Exanthema | interventions — Tooth Extraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — teeth and bone fragments of the jaw
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Normal tooth eruption
  Interventions: Procedure: Tooth extraction

INTERVENTIONS:
Procedure: Tooth extraction — Tooth extraction

SUMMARY:
The main objective is to study the expression of molecules involved in tooth morphogenesis and eruption in healthy patients, and then to compare them with the results in patients with abnormalities of eruption (results obtained via a collection of biological samples of rare diseases already authorized).

ELIGIBILITY:
Inclusion Criteria:

* Patient over 12 years old who has given his consent
* Patient whose legal representatives have given their consent for the use of operating waste destined for incineration
* Patient undergoing oral surgery at the University Hospitals of Strasbourg, at the origin of the production of surgical waste such as teeth and bone fragments
* Patient affiliated to a social security system

Exclusion Criteria:

* Refusal to participate
* Patient with chronic systemic pathology
* Patient under long-term drug treatment
* Patient presenting a rare pathology with oral manifestation
* Patient with a history of chemotherapy or head and neck radiotherapy
* Non-French speaking patient / inability to give informed information
* Patient under guardianship, curatorship or legal protection

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic (Hôpitaux Universitaires de Strasbourg, France)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Expression and localization of molecules involved in tooth eruption | During surgery
  Tissues are collected at the time of surgery and transferred during the day to the laboratory for analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided